CLINICAL TRIAL: NCT03303378
Title: Effects of Melatonin on Reperfusion Injury in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Effects of Melatonin on Reperfusion Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Wei Ren, MD, doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MelonRI
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Reperfusion Injury, Myocardial
Keywords: melatonin; Reperfusion Injury; myocardial infarction
MeSH Terms: conditions — Myocardial Reperfusion Injury; Reperfusion Injury; Myocardial Infarction | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Experimental): Patients will receive a total intravenous melatonin dose of 11.61 mg (aproximately 166 μg/kg).
  Interventions: Drug: melatonin (Helsinn Chemical Co, Biasca, Switzerland)
- Control group (Placebo Comparator): Patients will receive the same dose of placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: melatonin (Helsinn Chemical Co, Biasca, Switzerland) — Patients will receive a total intravenous melatonin (Helsinn Chemical Co, Biasca, Switzerland) dose of 11.61 mg (aproximately 166 μg/kg). The dose will be distributed in a volume of 500 ml of an isotonic and sterile solution of 100 μM melatonin during 150 min with a drip rate of 4.2 ml/min.
  The temporal distribution of perfusion will be: 30 min previous to percutaneous revascularization and remainder doses in a subsequent 120 min (1 h during the angioplasty +60 min post-intervention).
  Other Names: melatonin
  Arms: Melatonin group
Drug: Placebos — The temporal distribution of perfusion will be: 30 min previous to percutaneous revascularization and remainder doses in a subsequent 120 min (1 h during the angioplasty +60 min post-intervention).
  Other Names: Placebo
  Arms: Control group

SUMMARY:
Acute myocardial infarction is a major cause of mortality and morbidity. Primary percutaneous coronary intervention (pPCI) is currently the most effective treatment strategy in acute myocardial infarction. However, a sizable number of patients fail to restore optimal myocardial reperfusion, mostly because of the 'no-reflow' phenomenon. Melatonin is the chief indoleamine produced by the pineal gland, and a well-known antioxidant and free radical scavenger. Several studies have shown that melatonin protects against ischemia/reperfusion injury (IRI). In our previous study, melatonin markedly reduced infarcted area, improved cardiac function and reduced lactate dehydrogenase release in rats. The investigators planned to research the cardioprotective effects of intravenous melatonin administered prior to reperfusion and continued after restoration of coronary blood flow in patients with ST segment elevation myocardial infarction undergoing pPCI.

ELIGIBILITY:
Inclusion Criteria:

ST segment elevation myocardial infarction undergoing primary percutaneous poronary intervention

Exclusion Criteria:

* unconscious at presentation
* had cardiogenic shock
* had a history of myocardial infarction
* stent thrombosis
* renal insufficiency
* had previously undergone coronary artery bypass surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
The salvage index | 3 months after primary percutaneous coronary intervention
  The salvage index measured by cardiac magnetic resonance

SECONDARY OUTCOMES:
The final infarct size | 3 months after primary percutaneous coronary intervention
  The final infarct size measured by cardiac magnetic resonance
major adverse cardiovascular events (MACE) | 3 months after primary percutaneous coronary intervention
  recurrent myocardial infarction, recurrent angina, revascularization, heart failure, cardiac death.
treatment-emergent adverse events (TEAEs) | 3 months after primary percutaneous coronary intervention
  hypoglycemia, nausea

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dominguez-Rodriguez A, Abreu-Gonzalez P, de la Torre-Hernandez JM, Consuegra-Sanchez L, Piccolo R, Gonzalez-Gonzalez J, Garcia-Camarero T, Del Mar Garcia-Saiz M, Aldea-Perona A, Reiter RJ; MARIA Investigators. Usefulness of Early Treatment With Melatonin to Reduce Infarct Size in Patients With ST-Segment Elevation Myocardial Infarction Receiving Percutaneous Coronary Intervention (From the Melatonin Adjunct in the Acute Myocardial Infarction Treated With Angioplasty Trial). Am J Cardiol. 2017 Aug 15;120(4):522-526. doi: 10.1016/j.amjcard.2017.05.018. Epub 2017 May 30. PMID 28645475
- [Result] Zhou H, Zhang Y, Hu S, Shi C, Zhu P, Ma Q, Jin Q, Cao F, Tian F, Chen Y. Melatonin protects cardiac microvasculature against ischemia/reperfusion injury via suppression of mitochondrial fission-VDAC1-HK2-mPTP-mitophagy axis. J Pineal Res. 2017 Aug;63(1):e12413. doi: 10.1111/jpi.12413. Epub 2017 Apr 27. PMID 28398674
- [Result] Dominguez-Rodriguez A, Abreu-Gonzalez P, Garcia-Gonzalez MJ, Kaski JC, Reiter RJ, Jimenez-Sosa A. A unicenter, randomized, double-blind, parallel-group, placebo-controlled study of Melatonin as an Adjunct in patients with acute myocaRdial Infarction undergoing primary Angioplasty The Melatonin Adjunct in the acute myocaRdial Infarction treated with Angioplasty (MARIA) trial: study design and rationale. Contemp Clin Trials. 2007 Jul;28(4):532-9. doi: 10.1016/j.cct.2006.10.007. Epub 2006 Oct 17. PMID 17123867